CLINICAL TRIAL: NCT07405970
Title: A Phase 3 Clinical Study to Evaluate the Safety and Efficacy of Recombinant Humanized Monoclonal Antibody MIL62 Injection in the Treatment of Systemic Lupus Erythematosus.
Brief Title: A Phase 3 Clinical Study of MIL62 in Systemic Lupus Erythematosus
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Mabworks Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIL62-CT309
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIL62 (Experimental)
  Interventions: Drug: MIL62
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MIL62 — MIL62 will be administered by intravenous (IV) infusion at a dose of 1000 mg on Week (W) 1 Day (D) 1, W3D1, W25D1, W27D1.
  Arms: MIL62
Drug: Placebo — Placebo will be administered by intravenous (IV) infusion at a dose of 1000 mg on W1D1, W3D1, W25D1, W27D1.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of MIL62 compared with placebo in participants with systemic lupus erythematosus.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 ;
2. Diagnosis of systemic lupus erythematosus according to European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) SLE classification criteria ;
3. Positive antinuclear antibodies (ANA) ≥ 1:80 at screening or positive anti- dsDNA ;
4. High disease activity at screening ,SLEDAI-2000 score ≥8 (excluding alopecia score);
5. On a stable dose of one or more standard treatments for SLE prior to the first administration；
6. Able and willing to provide written informed consent and to comply with the study protocol.

Exclusion Criteria:

1. Unsufficient organ function;
2. Received rituximab or any B-cell depleting drug within 9 months prior to the first dose;
3. Subjects with CD4+ T lymphocyte count < 200 cells/μL;
4. Received cyclophosphamide within 8 weeks prior to the first dose; received calcineurin inhibitors (cyclosporine, tacrolimus, etc., except for topical use) or plasma exchange therapy within 4 weeks prior to the first dose;
5. Received a B-cell stimulating factor inhibitor such as Belimumab, and Telitacicept within 8 weeks prior to the first administration;
6. TNF inhibitor, interleukin monoclonal antibody, JAK inhibitor, BTK inhibitor, TYK2 inhibitor, or thalidomide within 4 weeks prior to the first administration;
7. Received live or attenuated vaccination within 28 days prior to the first administration;
8. Participated in other clinical trials within 28 days prior to the first administration;
9. Concomitant with other serious diseases;
10. Positive for hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb) with HBV DNA titer above the normal range; positive for hepatitis C virus (HCV) antibody; positive for human immunodeficiency virus (HIV);
11. Subjects with known history of severe allergic reactions to humanized monoclonal antibodies MIL62;
12. Breastfeeding or pregnant women;
13. Childbearing potential and unwillingness or impossibility to comply with a scientifically acceptable birth-control method;
14. Other conditions unsuitable for participation in this study determined by the Investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving SRI-4 at Week 52 | at Week 52

SECONDARY OUTCOMES:
Proportion of participants achieving SRI-4 at Week 24 | at Week 24
Changes in 24-hour urine protein in patients with baseline 24-hour urine protein elevation (24-hour urine protein ≥0.5g) at Week 24, 52 | at Week 24,52
Percentage of participants who achieved or maintained a prednisone dose of ≤7.5 mg/day (or equivalent dose) during Weeks 40 to 52 | from Week 40 to Week 52 after randomization
Change From Baseline in EuroQol- 5 Dimension (EQ-5D) at Week 24, 52 | up to 52 weeks after randomization
Change From Baseline in Serum Immunoglobulin Levels at Week 24 Change from baseline in the serum levels of IgG, IgA, IgM | up to 52 weeks after randomization
Change From Baseline in biomarkers associated with disease anti-dsDNA ,complement component 3 (C3), and complement component 4 (C4) | up to 52 weeks after randomization
Percentage of Participants with Adverse Events | up to 52 weeks after randomization
Pharmacodynamics(PD) characteristics: summarizing the changes in the absolute counts and percentages of peripheral blood CD19⁺ B cells | up to 52 weeks after randomization
Anti-Drug Antibodies (ADA) will be tested and percentage of ADA positive patients will be calculated to evaluate immunogenicity of MIL62 | up to 52 weeks after randomization

OTHER OUTCOMES:
Percentage of participants achieving Lupus Low Disease Activity State (LLDAS) at Week 52 | at Week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China